CLINICAL TRIAL: NCT05281848
Title: Evaluation of the Effect of Non-surgical Periodontal Treatment on Salivary and Gingival Crevicular Fluid Levels of IL-17 and IL-35 in Periodontitis Patients as Smoker and Non-smoker
Brief Title: Effect of Smoking and Periodontal Therapy on Salivary and Gingival Crevicular IL-17 and IL-35
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ezgi Sıla Taşkaldıran, Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21071282-050.99
Record Dates: First submitted 2020-03-02; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Periodontitis; Periodontal Diseases; Smoking; Smoking, Tobacco
Keywords: periodontitis; non-surgical periodontal treatment; IL-17; IL-35; saliva; gingival crevicular fluid
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Smoking; Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: A total of 55 subjects will be grouped as: 18 non-smoker patients with periodontitis (Group 1), 19 smoker patients with periodontitis (Group 2), 18 non-smoker and periodontally healthy individuals who will refer to our department. Spitting method will be used for collecting saliva samples. The paper strip method will be used for gingival crevicular fluid (GCF) sample collection. Samples will be taken from the mesial and distal surfaces of the teeth (healthy or have greater than or equal to 5mm pocket depth) after isolation from the saliva. Paper strips will be transferred to polypropylene tubes and stored at -30 ° C until inspection. After collecting samples, non-surgical periodontal treatment will be performed to all individuals which are classified as Group 1 and Group 2. Collection of saliva and GCF samples will be repeated at the 1st month after the end of treatment. ELISA kits will be used for the detection of saliva and GCF's IL-17 and IL-35.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Smoker-Periodontitis; Non-surgical periodontal treatment (Active Comparator)
  Interventions: Procedure: Non-surgical periodontal treatment
- Nonsmoker-Periodontitis;Non-surgical periodontal treatment (Active Comparator)
  Interventions: Procedure: Non-surgical periodontal treatment
- Healthy (No Intervention)

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Non-surgical periodontal treatment includes periodontal prophylaxis and root planning. No other methods or any of drugs will be used.
  Arms: Nonsmoker-Periodontitis;Non-surgical periodontal treatment; Smoker-Periodontitis; Non-surgical periodontal treatment

SUMMARY:
Periodontal diseases are among the major causes of tooth loss. Smoking may play a role as a contributing factor in the development of periodontitis by reducing the immune response. The role of cytokines in the pathogenesis of periodontal disease is clearly indicated in the literature; it has been shown that microorganisms that cause periodontal disease cause cytokine increase in saliva, gingival tissue and gingival crevicular fluid. Among these cytokines, interleukin (IL) -17 is proinflammatory and IL-35 is antiinflammatory and has been associated with periodontal disease.

DETAILED DESCRIPTION:
Periodontal diseases are among the complex inflammatory diseases that are considered among the leading causes of tooth loss, mostly observed with multiple etiological factors. The complexity of periodontal disease is due to the presence of the biofilm and the accompanying host response together.

Smoking, which is considered as one of the risk factors in terms of periodontitis, is one of the most preventable risk factors that affect the periodonium with many different mechanisms. Smoking plays a role in the etiopathogenesis of periodontitis, with its physiological changes in gingival tissue and its effects on host response and is considered to be an established risk factor. Although the effects of smoking on host response and its role in increasing the risk of periodontal disease are still being investigated, its effects on natural and acquired immune response cells have been studied separately. Consequently, components of cigarette suppress the immune system's defense responses; however, it has been reported to exacerbate pathological reactions.

The process of progression from periodontal health to periodontitis is formed by biofilm pathogens and host immune responses activated by these microorganisms. Intercellular communication is crucial during the progression of chronic inflammatory diseases, such as periodontitis. Cytokines, one of these ways of communication, are soluble proteins produced by various types of cells, such as structural and inflammatory cells, responsible for maintaining a complex network of communication between homotypic and heterotypic cell groups.

Interleukin-17 (IL-17) is a pro-inflammatory cytokine mostly stimulated from Th17 cells, stimulating inflammatory processes with many different mechanisms.

IL-35 inhibits the differentiation of Th17 cells and suppresses IL-17 production and therefore plays a protective role in Th17-related diseases.

There are many studies evaluating the effect of non-surgical periodontal treatment on individuals with smokers with periodontitis. However, the obtained results do not allow a clear data to be revealed. To exemplify, when the studies which investigates the evaluation of non-surgical periodontal treatment on IL-17 levels were evaluated, contradictory results were determined. In addition, as a result of our research, no studies evaluating the effects of non-surgical periodontal treatment on IL-35 levels in smokers with periodontitis have not been found.

ELIGIBILITY:
Inclusion Criteria:

* To be volunteer to participate in the study
* To be over 18
* Being systemically healthy
* Having greater than or equal to 15 teeth out of 3rd molar teeth
* To have localized or generalized periodontitis for the experimental group (clinical attachment loss in at least 6 surrounding areas and presence of greater than or equal to 5 mm periodontal pocket)
* For Smoking group; more than 10 cigarettes a day for more than 5 years
* For non-smokers; have not smoked for at least 3 years.

Exclusion Criteria:

* Have any systemic disease affecting periodontal condition
* To receive periodontal treatment in the last 6 months
* Use any medication that may affect the inflammatory process in the last 3 months
* Use local or systemic antibiotics in the last 3 months
* Pregnancy or lactation for female patients
* Regular use of mouthwash

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
IL-17 levels in gingival crevicular fluid | Change from baseline to 1st month after non-surgical periodontal treatment
  by ELISA method
IL-17 levels in saliva | Change from baseline to 1st month after non-surgical periodontal treatment
  by ELISA method
IL-35 levels in gingival crevicular fluid | Change from baseline to 1st month after non-surgical periodontal treatment
  by ELISA method
IL-35 levels in saliva | Change from baseline to 1st month after non-surgical periodontal treatment
  by ELISA method

SECONDARY OUTCOMES:
Plaque Index (PI) | Change from baseline to 1st month after non-surgical periodontal treatment
  by using Williams periodontal probe; Scores from 0 to 3, 0 is no visible plaque, 3 is visible plaque or dental calculus.
Gingival Index (GI) | Change from baseline to 1st month after non-surgical periodontal treatment
  by using Williams periodontal probe; Scores from 0 to 3, 0 is healthy gingiva, 3 is diseased gingiva with spontaneous bleeding.
Pocket Depth (PD) | Change from baseline to 1st month after non-surgical periodontal treatment
  by using Williams periodontal probe with milimeter signs; Pocket Depth is registered by milimeters.
Bleeding in Probing Index (BOP) | Change from baseline to 1st month after non-surgical periodontal treatment
  by using Williams periodontal probe; BOP is registered with + or - according to the presence of bleeding on probing.
Clinical Attachment Loss (CAL) | Change from baseline to 1st month after non-surgical periodontal treatment
  by using Williams periodontal probe with milimeter signs; CAL is registered by milimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Tüter, Professor, Study Director — Gazi University Dentistry Faculty Department of Periodontology
Locations (2):
- Turkey (Türkiye) (2):
  - Gazi University Faculty of Dentistry, Ankara
  - Gazi University Faculty of Medicine Immunology Department, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Page RC, Kornman KS. The pathogenesis of human periodontitis: an introduction. Periodontol 2000. 1997 Jun;14:9-11. doi: 10.1111/j.1600-0757.1997.tb00189.x. No abstract available. PMID 9567963
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S173-S182. doi: 10.1002/JPER.17-0721. PMID 29926951
- [Background] Kinane DF, Stathopoulou PG, Papapanou PN. Periodontal diseases. Nat Rev Dis Primers. 2017 Jun 22;3:17038. doi: 10.1038/nrdp.2017.38. PMID 28805207
- [Background] Page RC, Schroeder HE. Pathogenesis of inflammatory periodontal disease. A summary of current work. Lab Invest. 1976 Mar;34(3):235-49. PMID 765622
- [Background] Preshaw PM. Host modulation therapy with anti-inflammatory agents. Periodontol 2000. 2018 Feb;76(1):131-149. doi: 10.1111/prd.12148. Epub 2017 Nov 29. PMID 29193331
- [Background] Okada H, Murakami S. Cytokine expression in periodontal health and disease. Crit Rev Oral Biol Med. 1998;9(3):248-66. doi: 10.1177/10454411980090030101. PMID 9715365
- [Background] Zhang JM, An J. Cytokines, inflammation, and pain. Int Anesthesiol Clin. 2007 Spring;45(2):27-37. doi: 10.1097/AIA.0b013e318034194e. PMID 17426506
- [Result] Qiu F, Liang CL, Liu H, Zeng YQ, Hou S, Huang S, Lai X, Dai Z. Impacts of cigarette smoking on immune responsiveness: Up and down or upside down? Oncotarget. 2017 Jan 3;8(1):268-284. doi: 10.18632/oncotarget.13613. PMID 27902485
- [Result] Cua DJ, Tato CM. Innate IL-17-producing cells: the sentinels of the immune system. Nat Rev Immunol. 2010 Jul;10(7):479-89. doi: 10.1038/nri2800. Epub 2010 Jun 18. PMID 20559326
- [Result] Yao Z, Painter SL, Fanslow WC, Ulrich D, Macduff BM, Spriggs MK, Armitage RJ. Human IL-17: a novel cytokine derived from T cells. J Immunol. 1995 Dec 15;155(12):5483-6. PMID 7499828
- [Result] Vignali DA, Kuchroo VK. IL-12 family cytokines: immunological playmakers. Nat Immunol. 2012 Jul 19;13(8):722-8. doi: 10.1038/ni.2366. PMID 22814351
- [Result] Eshghipour B, Tofighi H, Nehal F, Vohra F, Javed F, Akram Z. Effect of scaling and root planing on gingival crevicular fluid cytokine/chemokine levels in smokers with chronic periodontitis: A systematic review. J Investig Clin Dent. 2018 Aug;9(3):e12327. doi: 10.1111/jicd.12327. Epub 2018 Feb 15. PMID 29450974
- [Derived] Ezgi Sila T, Gulay T, Aysegul AY, Melek Y. Non-surgical periodontal treatment effects on IL-17 and IL-35 levels in smokers and non-smokers with periodontitis. Odontology. 2025 Sep 19. doi: 10.1007/s10266-025-01207-0. Online ahead of print. PMID 40971113